CLINICAL TRIAL: NCT00001033
Title: The Treatment of Pulmonary Mycobacterium Tuberculosis in HIV Infection
Brief Title: The Treatment of Tuberculosis in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 222; CPCRA 019; 11199 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Isoniazid; Tuberculosis, Pulmonary; Pyrazinamide; Pyridoxine; Ofloxacin; Rifampin; AIDS-Related Opportunistic Infections; Ethambutol; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — HIV Infections; Tuberculosis; Tuberculosis, Pulmonary; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Ethambutol; Isoniazid; Pyrazinamide; Pyridoxine; Levofloxacin; Rifampin

INTERVENTIONS:
Drug: Ethambutol hydrochloride
Drug: Isoniazid
Drug: Pyrazinamide
Drug: Pyridoxine hydrochloride
Drug: Levofloxacin
Drug: Rifampin

SUMMARY:
PER 5/30/95 AMENDMENT: To compare the combined rate of failure during therapy and relapse after therapy between two durations of intermittent therapy (6 versus 9 months) for the treatment of pulmonary tuberculosis (TB) in HIV-infected patients. To compare toxicity, survival, and development of resistance in these two regimens.

ORIGINAL: To compare the efficacy and safety of induction and continuation therapies for the treatment of pulmonary TB in HIV-infected patients who are either from areas with known high rates of resistance to one or more anti-TB drugs or from areas where TB is expected to be susceptible to commonly used anti-TB drugs.

PER 5/30/95 AMENDMENT: In HIV-negative patients, intermittent anti-TB therapy has been shown to be as effective as daily therapy, but the optimal duration of therapy in HIV-infected patients has not been established.

ORIGINAL: In some areas of the country, resistance to one or more of the drugs commonly used to treat TB has emerged. Thus, the need to test regimens containing a new drug exists. Furthermore, the optimal duration of anti-TB therapy for HIV-infected patients with TB needs to be determined.

DETAILED DESCRIPTION:
PER 5/30/95 AMENDMENT: In HIV-negative patients, intermittent anti-TB therapy has been shown to be as effective as daily therapy, but the optimal duration of therapy in HIV-infected patients has not been established.

ORIGINAL: In some areas of the country, resistance to one or more of the drugs commonly used to treat TB has emerged. Thus, the need to test regimens containing a new drug exists. Furthermore, the optimal duration of anti-TB therapy for HIV-infected patients with TB needs to be determined.

PER 5/30/95 AMENDMENT: Patients who have received an acceptable induction regimen prior to study entry and have been found to be susceptible to isoniazid and rifampin with no pyrazinamide resistance are randomized to receive either isoniazid or rifampin plus vitamin B6 biweekly for 18 or 31 weeks. Patients are evaluated at months 1, 2, 4, 6, 8, and 10, and every 4 months thereafter. Minimum follow-up is 1.5 years.

ORIGINAL: In the induction phase, patients enrolled in "drug-susceptible" areas (defined as metropolitan areas with a resistance rate for isoniazid therapy of less than 10 percent) receive four drugs: isoniazid (plus pyridoxine), rifampin, pyrazinamide, and ethambutol. Patients enrolled in "drug-resistant" areas (resistance rate for isoniazid of 10 percent or higher) receive the four-drug regimen with or without a fifth drug, levofloxacin. After 8 weeks of induction, patients with multi-drug resistance are removed from study regimens; all other patients enter a continuation phase. Pansusceptible patients (showing susceptibility to all first-line anti-TB drugs) receive two study drugs for an additional 18 or 31 weeks; patients with isoniazid-resistant (or intolerant) TB receive two or three study drugs for an additional 44 weeks, while those with rifampin-resistant TB receive two or three study drugs for an additional 70 weeks. Patients are evaluated every 2 weeks in the induction phase and every 12 weeks in the continuation phase. Minimum follow-up is 2 years.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

INDUCTION PHASE (ELIMINATED PER 5/30/95 AMENDMENT).

* HIV infection.
* Diagnosis of pulmonary TB.

NOTE:

* Patients from "susceptible" areas may be 13 years of age or older. Patients from "resistant" areas must be 18 years of age or older.

CONTINUATION PHASE.

* Successful completion of induction phase and confirmation of TB by culture and susceptibility results.
* Susceptibility to and tolerance of isoniazid and rifampin and no resistance to pyrazinamide.
* HIV infection.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Multi-drug resistance to at least isoniazid and rifampin or known to have had close contact with a person with known multi-drug resistant TB.
* Known treatment-limiting reaction to any of the study drugs.
* Other disorders or conditions for which the study drugs are contraindicated.

Concurrent Medication:

Excluded:

* Other medications with anti-TB activity.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650
Dates: Study Completion 1997-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perlman D, Study Chair; El-Sadr W, Study Chair
Locations (12):
- United States (12):
  - USC CRS, Los Angeles, California
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - SUNY - Buffalo, Erie County Medical Ctr, Buffalo, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Telzak EE, Chirgwin K, Nelson E, Matts J, Benson C, Sepkowitz K, Perlman D, El-Sadr W. Predictors for multidrug-resistant tuberculosis (MDRTB) among HIV-infected patients and response to specific MDRTB drug regimens. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:184 (abstract no 647)
- [Background] el-Sadr WM, Perlman DC, Matts JP, Nelson ET, Cohn DL, Salomon N, Olibrice M, Medard F, Chirgwin KD, Mildvan D, Jones BE, Telzak EE, Klein O, Heifets L, Hafner R. Evaluation of an intensive intermittent-induction regimen and duration of short-course treatment for human immunodeficiency virus-related pulmonary tuberculosis. Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA) and the AIDS Clinical Trials Group (ACTG). Clin Infect Dis. 1998 May;26(5):1148-58. doi: 10.1086/520275. PMID 9597244
- [Background] Perlman DC, el-Sadr WM, Nelson ET, Matts JP, Telzak EE, Salomon N, Chirgwin K, Hafner R. Variation of chest radiographic patterns in pulmonary tuberculosis by degree of human immunodeficiency virus-related immunosuppression. The Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA). The AIDS Clinical Trials Group (ACTG). Clin Infect Dis. 1997 Aug;25(2):242-6. doi: 10.1086/514546. PMID 9332519
- [Background] Perlman DC, El Sadr WM, Heifets LB, Nelson ET, Matts JP, Chirgwin K, Salomon N, Telzak EE, Klein O, Kreiswirth BN, Musser JM, Hafner R. Susceptibility to levofloxacin of Myocobacterium tuberculosis isolates from patients with HIV-related tuberculosis and characterization of a strain with levofloxacin monoresistance. Community Programs for Clinical Research on AIDS 019 and the AIDS Clinical Trials Group 222 Protocol Team. AIDS. 1997 Oct;11(12):1473-8. doi: 10.1097/00002030-199712000-00011. PMID 9342069